CLINICAL TRIAL: NCT04469205
Title: Randomized and Prospective Study to Assess the Impact of Personalized Coaching on the Time Period and Quality of Return to Work After Breast Cancer
Brief Title: Study to Assess the Impact of Personalized Coaching on the Time Period and Quality of Return to Work After Breast Cancer
Acronym: OPTICOACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruiting
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IC 2017-06
Record Dates: First submitted 2020-06-08; First posted 2020-07-13 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): intervention group that will receive return-to-work coaching sessions. The intervention consists of 3 individual coaching sessions with a certified professional coach. This personalized accompaniment will complete the standard accompaniment offered to all patients.
  Interventions: Other: Coaching sessions
- Control Group (No Intervention): control group who will receive the current care which consists of a psychosocial care.
  This care consists in offering the patient regular information meetings organized with social workers of the Health Insurance, to consult a psychologist and to access patients' homes at the frequency of their choice and according to their need.

INTERVENTIONS:
Other: Coaching sessions — There are 3 sessions : the first session will last 1h30 and will be in consultation within the Institut Curie. The second session will last 1h30 and will be done remotely (by phone or by videoconference). The duration of the 3rd and last session will be adapted according to the needs of each patient and will last a maximum of 1 hour. It will also be done remotely (by phone or by videoconference).
  Arms: Intervention Group

SUMMARY:
Evaluate the impact of coaching sessions on the return to work rate (number of patients returning at work / total number of patients per arm) 6 months after inclusion in the study for breast cancer in professionnally active patients.

ELIGIBILITY:
Inclusion Criteria:

Any patient active at the time of the diagnosis of breast cancer, treated consecutively at the Institut Curie during the study period, and whose first treatment will be surgery, will be offered participation in the study.

1. Invasive non-metastatic breast cancer, treated first by surgery
2. Age ≥ 18 and ≤ 60 years
3. Active woman at the time of diagnosis
4. Patient with internet access and email address
5. Patient affiliated with a social security scheme, speaking and reading French
6. Signature of informed consent

Exclusion Criteria:

1. In situ breast cancer
2. History of breast cancer
3. Metastatic breast cancer
4. Inflammatory Breast Cancer
5. Woman with a life expectancy <6 months at the time of diagnosis (in relation to other serious chronic diseases)
6. Persons deprived of liberty or under guardianship
7. Impossibility to submit to the medical follow-up of the test for geographical, social or psychological reasons

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Impact of coaching sessions on the return to work rate (number of patients returning at work / total number of patients per arm) 6 months after inclusion in the study | 6 months
  The rate of patients returning to work (part-time or full-time) for more than 2 weeks to 6 months of inclusion in the study in each group.

SECONDARY OUTCOMES:
Quality of the return to work | 6 and 12 months
  Evaluation of the quality of the return to work at 6 and 12 months after inclusion by questionnaire VOW / QFT (in case of return to work only).
  Evaluation scale : 1=never to 4=ever
Sustainability of the return to work | 6 and 12 months
  Evaluation of the durability of the return to work at 6 and 12 months after inclusion by registration by the patients of the number of days off work and / or working time arrangement
Impact of the return to work / work stoppage on the quality of life | 6 and 12 months
  Evaluation of the impact of return to work / work stoppage on the quality of life estimated by QLQ-C30 questionnaire at baseline and at 6 and 12 months post-inclusion
The production losses related to presenteeism during maintenance or return to work | 6 and 12 months
  Evaluation of production losses related to presenteeism at the time of maintenance or return to work at 6 and 12 months post inclusion, by collecting the number of days worked during the study period (12 months)
The production losses related to presenteeism during maintenance or return to work | 6 and 12 months
  Evaluation of the loss of productivity during a professional activity : in case of return to work, the "Work limitation questionnaire" will be completed at 6 and 12 months after inclusion
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 12 months
  Determining the determinants of return to work at 6 and 12 months post inclusion using the QLQ-BR23questionnaire.
  Evaluation scale : 0=not at all to 4=a lot
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 6 and 12 months
  Determining the determinants of return to work at 6 and 12 months post inclusion using the QLQ-FA12 questionnaire.
  Evaluation scale : 0=not at all to 4=a lot
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 6 and 12 months
  Determining the determinants of return to work at 6 and 12 months post inclusion using the HADS questionnaire.
  Anxiety scale : 3=most of the time to 0=never Depression scale : 3=never to 0= most of the time
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 6 and 12 months
  Determining the determinants of return to work at 6 and 12 months post inclusion using the SSQ6 questionnaire.
  Evaluation scale : 1=really dissatisfied to 6 =really satisfied
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 6 and 12 months
  Determining the determinants of return to work at 6 and 12 months post inclusion using the Brief Cope questionnaire.
  Evaluation scale : 0=not at all to 4=absolutely
The determinants of return to work (factors associated with a return to work "successful": early, sustainable and quality) | 6 and 12 months
  These determinants will also be evaluated through the collection of socio-demographic data, cancer characteristics and treatments administered.
The medico-economic impact of returning to work | 12 months
  Evaluation of the medico-economic impact of return to work by comparing the costs of care in the two groups

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).